CLINICAL TRIAL: NCT03657940
Title: Impact of a Multicomponent Exercise Program (VIVIFRAIL)on Functional Capacity in Frail Community Aged Participants With Cognitive Decline . Multi-center Randomized Control Trial
Brief Title: Impact of a Multicomponent Exercise Program on Functional Capacity in Frail Aged Participants With Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Matia Foundation (Other); Hospital Universitario Getafe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Gov NA 28-16
Record Dates: First submitted 2018-07-30; First posted 2018-09-05 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Frail Elderly Syndrome; Cognitive Impairment
Keywords: Exercise therapy
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise intervention (Experimental): multicomponent exercise training program [VIVIFRAIL],
  Interventions: Behavioral: VIVIFRAIL multicomponent exercise training program
- Usual Care (No Intervention): Participants randomly assigned to the usual care group will receive normal outpatient care, which includes physical rehabilitation when needed.

INTERVENTIONS:
Behavioral: VIVIFRAIL multicomponent exercise training program — The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individual's functional capacity, using dumbbells aiming for 2-3 sets of 10-15 repetitions at an intensity of 30-50% of 1Repetition Maximum ( combined with balance-training, flexibility and gait exercises that progressed in difficulty.
  Arms: Exercise intervention

SUMMARY:
Randomized Controlled trial of 370 aged participants over 75 years old coming from clinics of Geriatric Departments in three University Hospitals in Spain (Pamplona, Getafe y San Sebastián). Participants who met inclusion criteria will be randomized to control (usual care)l or intervention group (multicomponent exercise program). The main objective of the trial is to study the effect of a multicomponent exercise training program (resistance, aerobic, strength, balance and flexibility) in frail aged participants who live in the community with cognitive decline in: functional capacity, strength, power, cognition, falls , depression, quality of life, institutionalization and hospital admissions

DETAILED DESCRIPTION:
Usual care group (control) Participants randomly assigned to the usual care group will receive normal outpatient care, which includes physical rehabilitation when needed.

Intervention group (training) The intervention will consist of a multicomponent exercise training programme -VIVIFRAIL-(A Practical Guide for Prescribing a Multi-Component Physical Training Program to prevent weakness and falls in People over 70, Showed in www.vivifrail.com), which will be composed of supervised progressive resistance training, balance-training, flexibility and cardiovascular for 7 days/week. During the training period, patients will be trained between 2 and 120 minutes each day.

The supervised multicomponent exercise training programme will be comprised of upper and lower body strengthening exercises, tailored to the individual's functional capacity, using dumbbells aiming for 2-3 sets of 10-15 repetitions at an intensity of 30-50% of 1RM combined with balance-training, flexibility and gait exercises that progressed in difficulty. The resistance exercises focused on the major upper and lower limb muscles. During the progressive resistance training, instruction will be provided to the participants to perform the exercises at a high velocity of motion. However, care will be taken to ensure that exercises were executed with correct form. Balance and gait training exercises that progressed in difficulty will be also implemented: e.g. semitandem foot standing, line walking, stepping practice, walking with small obstacles, proprioceptive exercises, and altering the base of support and weight transfer from one leg to the other. An experienced physical trainer will carefully explain all the exercises. Participants and their carer / family members will be carefully familiarized with the training procedures in advance.

ELIGIBILITY:
Inclusion Criteria:

* - Age: 75 years or older.
* Able to ambulate with or without personal/technical assistance.
* Barthel Index ≥ 60.
* Able to communicate.
* Mild cognitive impairment or Dementia level GDS-4.
* Fragility o pre-frailty according to Linda Fried ≥ 1.
* Subjects should have someone to help them do the exercises.
* Informed consent: Must be capable and willing to provide consent.

Exclusion Criteria:

* Any factor precluding performance of the physical training programme or testing procedures as determined by the attending physician. These factors include, but are not limited to the following:
* Myocardial infarction in the past 3 months.
* Unstable Angina pectoris.
* Terminal illness.
* Uncontrolled arrhythmia.
* Unstable cardiovascular disease or other medical condition.
* Uncontrolled arterial hypertension.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Changes from baseline to 1st and 3th months of follow up
  The functional capacity of patients will be evaluated by the Short Physical Performance Battery (SPPB) which evaluates, balance, gait ability, and leg strength using a single tool. The total score ranges from 0 (worst) to 12 points (best). The SPPB test has been shown to be a valid instrument for screening frailty and predicting disability, institutionalization, and mortality. A total score of less than 10 indicates frailty and a high risk of disability and falls. A one-point change in the score has clinical relevance

SECONDARY OUTCOMES:
Barthel index | Changes from baseline to 1st and 3th months of follow up
  international and validated tool of disability. The score range from 0 (severe functional dependence) to 100 (functional independence
Handgrip strength in the dominant hand | Changes from baseline to 1st and 3th months of follow up
  Loss of handgrip strength in the dominant hand evaluated with a dynamometer is a useful tool for the measurement of functional capacity. This characteristic is a strong predictor of disability, morbidity, and mortality as well as one of the components of Fried's frailty phenotype. Higher values indicates better function Ranges of normality are corrected by BMI. For example for men with a BMI less of 24 , normality is consider over 29 kg
6-metre gait velocity test (GVT). | Changes from baseline to 1st and 3th months of follow up
  Gait ability will be assessed using the 6-metre gait velocity test (GVT). Starting and ending limits will be marked on the floor with tapelines for a total distance of 8 meters. Participants will be instructed to walk in their self-selected usual pace for two attempts. The best result of both trials will be registered. The first and last metre, considered the warm-up and deceleration phases, respectively, will not be included in calculations of the gait assessment. Higher scores ( > 1.0 m/s) indicates better functional capacity and lower scores (< 0.8 m/s) scores worse functional capacity
MEC-Lobo cognitive test | Changes form baseline to 1st and 3th months of follow up
  cognitive function will be measured will the Spanish Version of MMSE ( MEC-Lobo) in case of dementia. It ranges from 0 ( worse score ) to 35 (best score). A score less than 23 indicates significative cognitive decline
MOCA( Montreal Cognitive Assessment) test | Changes from baseline to 1st and 3th months of follow up
  cognitive function will be measured with MOCA ( Montreal Cognitive Assessment Test) in case of mild cognitive decline. The MOCA is a validated test in Spanish It ranges from 0 ( worse score ) to 30 (best score). A score less than 26 indicates suggest mild cognitive decline
Trail Making Test part A ( TMT-A) | Changes from baseline to 1st and 3th months of follow up
  Executive function will be assessed with the Trail Making Test part A. Results for TMT A are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.Average will be consider 29 seconds, Deficient > 78 seconds and Rule of Thumb most 90 seconds.
Isometric lower limb strength test (right knee extensors and hip flexors) | Changes from baseline to 1st and 3th months of follow up
  Isometric lower limb (right knee extensors and hip flexors) muscle strength will be measured using a manual dynamometer. Higher values indicates better functional capacity
1Repetition Maximum (RM) Maximal dynamic strength test | Changes from baseline to 1st and 3th months of follow up
  Maximal dynamic strength will be assessed using the 1Repetition Maximum (RM) test in the bilateral leg press exercise using exercise machines (Exercycle, S.L., BH Group, Vitoria, Spain). In the first assessment, the subjects will warm up with specific movements for the exercise test. Each subject's maximal load will be determined in no more than five attempts, with a 3-min recovery period between attempts.
Repetitions at maximal velocity at intensities of 50% of 1RM test | Changes from baseline to 1st and 3th months of follow up
  Participants will perform ten repetitions at maximal velocity at intensities of 50% of 1RM to determine the maximum power (w) and the loss of power during the ten repetitions in the leg press exercise.Higher values indicates better functional capacity
Geriatric Depression Scale ( GDS) Yesavage abbreviated scale | Changes from baseline to 1st and 3th months of follow up
  Depression will be assessed wit the GDS Yesavage abbreviated scale of 15 items. Is is ranged between 0 ( best value) to 15 ( worse value). Scores between 0-5 indicates normality, 5-9 minor depression and scores over 9 indicates mayor depression
Categorical pain scale | Changes from baseline to and 3th months of follow up
  Pain will be assessed with a subjective categorical pain scale. It is ranged in four categories : 0 ( no pain), 4 ( litle bit), 6 ( quite) , 10 ( a lot)
Rate of falls | Baseline, 1st and 3th months of follow up
  Rate of new falls during follow up
Vivifrail risk of falls scale | Changes from baseline to 1st and 3th months of follow up
  Risk of falls will be assessed using Vivifrail methodology. High risk of falls is considered if one of the following questions is positive: 2 o more falls in the last year, a previous fall with medical attention and if the participant scores over 20 seconds in the time up and go test, TUG test ( time of rising from a chair, walking three meters and going back to sitting position) or less than 0.8 m/s in the Gait velocity test
Mortality | Changes from baseline to 1st and 3th months of follow up
  Mortality will be assessed with a clinical questionnaire during follow up.
Admissions to the hospital | Baseline, 1st and 3th months of follow up
  New admissions to the hospital will be assessed with a clinical questionnaire during follow up
Incidence of institutionalization to nursing homes | Baseline, 1st and 3th months of follow up
  New institutionalizations to nursing homes will be assessed with clinical questionary during follow up
Visit to emergency room | Baseline, 1st and 3th months of follow up
  Visits to emergency room will be assessed with a clinical questionnaire during follow up
Number of total Drugs | Changes from baseline to 3th month´s follow up
  Number of drugs during follow up will be assessed with a clinical questionnaire
Presence of 5 or more drugs ( Polypharmacy ) registration | Changes from baseline to 3th month´s follow up
  Registration of the presence of 5 or more drugs( Polypharmacy ) during follow -up will be done with a clinical questionnaire .
Psychotropic drugs (neuroleptics , cholinesterase inhibitors , antidepressants , benzodiazepines , anti-epileptics) registration | Changes from baseline to 3th month´s follow up
  Registration of the following physchotropic drugs will be assessed with a clinical questionnaire : neuroleptics , cholinesterase inhibitors , antidepressants , benzodiazepines , anti-epileptics
Neuropsychiatric Inventory Questionary (NPI) | Changes from baseline and 3th month´s follow up
  Assessment of psycho-behavioral symptoms associated to mild cognitive decline or dementia will be assessed with the Neuropsychiatric Inventory Questionary (NPI). NPI is a validated informant-based interview that assesses 12 neuropsychiatric symptoms over the previous month.Initial responses to each domain question are "Yes" (present) or "No" (absent). If the response to the domain question is "No", the informant goes to the next question. If "Yes", the informant then rates both the Severity of the symptoms present within the last month on a 3-point scale and the associated impact of the symptom manifestations on them (i.e. Caregiver distress) using a 5-point scale. The NPI provides symptom Severity and Distress ratings for each symptom reported, and total Severity and Distress scores reflecting the sum of individual domain scores.
Dual task gait ( arithmetic) 6 m velocity test | Changes from baseline to 1st and 3th months of follow up
  The dual-task paradigm will be used in the 6-m habitual GVT. Two trials will be conducted (best record will be taking in account) During the arithmetic dual-task condition (arithmetic GVT), we will assess gait velocity while participants are counting backward aloud from 100 by ones
Dual task gait (verbal) 6 m velocity test | Changes from baseline to 1st and 3th months of follow up
  The dual-task paradigm will be used in the 6-m habitual GVT. Two trials will be conducted(best record will be taking in account)During the verbal dual-task condition (verbal GVT), we will assess gait velocity while participants are naming animals by loud
EuroQol-5D (EQ-5D) quality of life assessment test | Changes from baseline to 3th month´s follow up
  Quality of of life will be assessed with an international validated scale EuroQol-5D (EQ-5D). Its composed by. It asses health status (mobility, personal care, basic and instrumental daily living activities , pain and ansiety/depression) ranged from 0 ( worst health status) to 100 ( best health status )
Registration of other geriatric syndromes (visual and hear impairment, urinary and fecal incontinence, delirium , dysphagia, constipation , pressure ulcers ) | Changes from baseline to 3th month´s follow up
  Presence of other geriatric syndromes ( visual and hear impairment, urinary and fecal incontinence, delirium , dysphagia, constipation , pressure ulcers ) will be assessed with a clinical questionnaire

OTHER OUTCOMES:
Mini- Nutritional Assessment (MNA) | Baseline visit
  The MNA® in the short form (MNA-SF) is a validated nutrition screening and assessment tool that can identify geriatric patients age 65 and above who are malnourished or at risk of malnutrition. Is is ranged from 0 to 14. 12-14 points indicates normal nutritional status : 8-11 points: At risk of malnutrition 0-7 points: Malnourished
Cumulative Illness Rating Scale for Geriatrics (CIRS-G) | Baseline visit
  This scoring system measures the chronic medical illness ("morbidity") burden while taking into consideration the severity of chronic diseases in 14 items representing individual body systems. The general rules for severity rating are:
  0→No problem affecting that system.
  1. Current mild problem or past significant problem.
  2. Moderate disability or morbidity and/or requires first line therapy.
  3. Severe problem and/or constant and significant disability and/or hard to control chronic problems.
  4. Extremely severe problem and/or immediate treatment required and/or organ failure and/or severe functional impairment.
  The cumulative final score can vary theoretically vary from 0 to 56 (although a very high score is impossible).
Functional Activities Questionnaire (FAQ) | Changes from baseline to 1st and 3th months follow up
  The Functional Activities Questionnaire (FAQ) measures instrumental activities of daily living (IADLs), such as preparing balanced meals and managing personal finances. Since functional changes are noted earlier in the dementia process with IADLs that require a higher cognitive ability compared to basic activities of daily living (ADLs), this tool is useful to monitor these functional changes over time. It evaluates 10 items and it is necessary to ask informant to rate patient's ability using the following scoring system: • Dependent = 3
  * Requires assistance = 2
  * Has difficulty but does by self = 1
  * Normal = 0
  * Never did [the activity] but could do now = 0
  * Never did and would have difficulty now = 1 It is ranged between 0-30. Cut-point of 9 (dependent in 3 or more activities) is recommended to indicate impaired function and possible cognitive impairment.
Isaacs set test | Changes from baseline to 3th month´s follow up
  The set test is a simple rapid test of mental function which requires the subject to recall items form different common categories. In our case we choose a fluency verbal test because it´s simplicity in participants with sensorial deficits and illiteracy . We will ask the participants to say by loud in one minute words that starts with word "P". correct and wrong answers will be noted. More words indicates better cognitive function
Gait regularity analysis with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait regularity analysis will be performed
Gait cadence analysis with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait cadence analysis will be performed
Gait variability analysis with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait variability analysis will be performed
Gait symmetry analysis with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional tasks (such as balance, gait and rising form a chair ) and cognitive evaluations (dual tasking), an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Gait symmetry analysis will be performed
Five Times Sit to Stand peak power analysis test with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Peak power analysis will be performed
Five Times Sit to Stand impulse analysis test with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Impulse analysis will be performed
Five Times Sit to Stand orientation analysis test with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional Five Times to Stand Test an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Orientation analysis will be performed
Balance power spectrum analysis test with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional balance assessment an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Power spectrum analysis will be performed
Balance area analysis test with an inertial sensor unit | Changes from baseline to 1st and 3th months follow up
  During functional balance assessment an inertial sensor unit (IU) will be attached over the lumbar spine (L3) to record the acceleration data in control and intervention participants. Balance area analysis will be performed

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Casas Herrero, MD PhD, Principal Investigator — Complejo Hospitalario de Navarra/Fundación Navarrabiomed
Locations (1):
- Fundación Miguel Servet/ Navarrabiomed, Pamplona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Casas-Herrero A, Saez de Asteasu ML, Anton-Rodrigo I, Sanchez-Sanchez JL, Montero-Odasso M, Marin-Epelde I, Ramon-Espinoza F, Zambom-Ferraresi F, Petidier-Torregrosa R, Elexpuru-Estomba J, Alvarez-Bustos A, Galbete A, Martinez-Velilla N, Izquierdo M. Effects of Vivifrail multicomponent intervention on functional capacity: a multicentre, randomized controlled trial. J Cachexia Sarcopenia Muscle. 2022 Apr;13(2):884-893. doi: 10.1002/jcsm.12925. Epub 2022 Feb 11. PMID 35150086
- [Derived] Casas-Herrero A, Anton-Rodrigo I, Zambom-Ferraresi F, Saez de Asteasu ML, Martinez-Velilla N, Elexpuru-Estomba J, Marin-Epelde I, Ramon-Espinoza F, Petidier-Torregrosa R, Sanchez-Sanchez JL, Ibanez B, Izquierdo M. Effect of a multicomponent exercise programme (VIVIFRAIL) on functional capacity in frail community elders with cognitive decline: study protocol for a randomized multicentre control trial. Trials. 2019 Jun 17;20(1):362. doi: 10.1186/s13063-019-3426-0. PMID 31208471